CLINICAL TRIAL: NCT01390467
Title: Cognitive Impact of Paracetamol in Healthy Volunteers
Acronym: ICP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0095; 2011-000662-35 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Paracetamol; Cognitive impact
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Cantab® — Randomized study, double-blind, crossover, controlled versus placebo.

SUMMARY:
Randomized study, double-blind, crossover, controlled versus placebo.

DETAILED DESCRIPTION:
Paracetamol impact on cognitive processes has been until recently little studied in literature that presents conflicting results. Some authors do not describe any cognitive performance change (Bradley and Nicholson, 1987) but more recent studies (Ishida et al., 2007) report an interesting performance improvement in therapeutic doses of paracetamol.

This improved performance would use the serotonergic pathway that is involved in the analgesic mechanism of paracetamol as the investigators demonstrated in our laboratory on previous work (Pickering et al. 2006, 2008). However, non-therapeutic dose, instead, showed a deterioration of memory processes in animals which may be link to implication of Cyclooxygenases COX-2. Indeed, several studies have demonstrated (Sharifzadeh et al. 2005; Teather et al., 2005) that anti COX-2 (such as Celebrex) cause in animal a deleterious effect on memory, while an anti COX1 and 2 (as indomethacin) or an anti COX1 (as piroxicam) lead to no change. A dose-effect relationship is therefore suggested on animals. Furthermore, a recent study in healthy volunteers showed that paracetamol acts not only on pain but also on pain / stress in society in everyday life (" social pain ") (deWall et al., 2010). By fMRI, these psychologists have shown that the reduction of "social" pain is associated with a decrease in neuronal activity in brain regions that are involved in social processes but also those who are involved in pain processes (anterior cingulate cortex , anterior insula etc..). They also showed that paracetamol known for its painkillers properties may reduce the painful feelings of rejection or shelved in everyday life. The cognitive-emotional impact of paracetamol is even more interesting that the investigators now know that its metabolism could involve cannabinoids receptors, particularly CB1 in hippocampus and association cortex involved themselves in cognitive phenomena.

INSERM U766 team to which the investigators belong has proposed the following sequence from preclinical : 1) metabolism of acetaminophen in analgesic metabolite AM404 via FAAH enzyme, 2) AM404 acts indirectly on CB1 receptors, 3) strengthening of bulbo spinal descending pathways by the endocannabinoid system, 4) involvement of serotonergic receptors pain suppressors.

This protocol follows a pilot that the investigators completed (HOP clinicaltrial.gov NCT01053650, unpublished results yet) where the investigators studied the impact of 2g of paracetamol in healthy volunteers. The investigators showed a memory improvement, but with no placebo group, it has not been possible to conclude a significant impact of oral paracetamol. Thus, this protocol will allow us to better understand if paracetamol can affect some cognitive processes, particularly vigilance, memory and decision making.

In addition, the investigators will build a biological collection to assess the pharmacogenetic profile of subjects and, in a secondary objective, correlate it to cognitive characteristics of subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers,
* aged over 18 years and not more than 25 years,
* males,
* free from any treatment in the 7 days preceding inclusion especially no use of analgesics or anti-inflammatories

Exclusion Criteria:

* Contraindications to the administration of paracetamol
* medical and/or surgical history judged by the investigator or his representative as being incompatible with the test, especially subjects with neuropathic pain
* evolutionary pathology at review for inclusion
* excessive intake of alcohol, tobacco (more than 10 cigarettes / day), coffee, tea or drinks containing caffeine (equivalent to more than 4 cups per day) or drug

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Assess cognitive impact of taking paracetamol within healthy volunteers by comparing the results on cognitive tests Cantab® between two passages, in particular a memory test (SOC) | after the results on cognitive tests Cantab

SECONDARY OUTCOMES:
Assess cognitive impact of taking paracetamol on other cognitive tests Cantab® (understanding : MOT and DMS, reaction time : RTI, visual memory : PRM, decision making : IST) | after an other cognitive test Cantab

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand